CLINICAL TRIAL: NCT03004742
Title: Influence of Ingesting a Flavonoid-rich Supplement on the Human Metabolome and Concentration of Urine Phenolics
Brief Title: Flavonoid-rich Supplement Influence on the Human Metabolome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: Reoxcyn Discoveries Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-0274
Record Dates: First submitted 2016-12-13; First posted 2016-12-29 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Inflammation
Keywords: polyphenols; metabolomics; oxidative stress
MeSH Terms: conditions — Inflammation | interventions — Flavonoids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flavonoid (Experimental): Flavonoid supplement
  Interventions: Dietary Supplement: Flavonoid
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Flavonoid — Flavonoid rich supplement
  Arms: Flavonoid
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will measure the effect of ingesting a flavonoid-rich supplement on various biomarkers in overweight/obese women during a 12-week period. The flavonoid-rich supplement contains a mixture of flavonoids including quercetin, catechins from green tea extract, and anthocyanins from bilberry extract, and other food components that facilitate flavonoid bioactivity including fish oil, caffeine, and vitamin C.

DETAILED DESCRIPTION:
1. The primary objective of this study is to evaluate the effect of ingesting a flavonoid-rich supplement on total urine polyphenol concentration and shifts in blood metabolites related to flavonoid intake in healthy but overweight/obese community-dwelling adults.
2. Secondary objectives are to determine related effects on measures of inflammation and oxidative stress. Studies are mixed regarding the influence of flavonoid supplements on traditional biomarkers for inflammation and oxidative stress, and metabolite shifts from the metabolomics measurements may provide better insights. Chemistry profiles and symptom logs will be compared pre- and post-study between groups to confirm prior safety data collected on human participants.

Hypothesis: Subjects randomized to ingestion of the flavonoid-rich supplement compared to placebo will experience an increase in total urine polyphenols concentrations and shifts in blood metabolites related to increased flavonoid metabolism. Secondarily, subjects ingesting the flavonoid-rich supplement will experience a decrease in systemic inflammation and oxidative stress.

BASELINE TESTING (ASU-NCRC HUMAN PERFORMANCE LAB):

A. One week before the start of the study, subjects will report to the ASU-NCRC Human Performance Lab, be oriented to the study, and provide voluntary consent. Subjects will fill in a medical health questionnaire to verify medical history and lifestyle habits. Subjects must agree to maintain normal dietary and physical activity patterns during the 12-week intervention, and not make formal attempts to lose body weight. All other subject inclusion and exclusion criteria must be maintained during the study. Subjects will be instructed on how to record all food intake during a 3-day period prior to the start of the study (Thursday, Friday, and Sunday).

Subjects will be instructed on how to collect urine for 24-hours during the day just before the study starts. Urine collection guidelines:

* You should collect every drop of urine during each 24-hour period. It does not matter how much or little urine is passed each time, as long as every drop is collected.
* Begin the urine collection in the morning after you wake up, after you have emptied your bladder for the first time.
* Urinate (empty the bladder) for the first time and flush it down the toilet. Note the exact time (eg, 6:15 AM). You will begin the urine collection at this time.
* Collect every drop of urine during the day and night in an empty collection bottle. Store the bottle in the refrigerator. Be sure to collect any urine passed during bowel movements.
* Finish by collecting the first urine passed the next morning, adding it to the collection bottle. This should be within ten minutes before or after the time of the first morning void on the first day (which was flushed). In this example, you would try to void between 6:05 and 6:25 on the second day. If you need to urinate one hour before the final collection time, drink a full glass of water so that you can void again at the appropriate time. If you have to urinate 20 minutes before, try to hold the urine until the proper time.
* Please note the exact time of the final collection.

B. On the first day of the study, subjects will return to the lab in a fasted state (9 or more hours with no food or beverage other than water) and turn in the 3-day food record and the 24-h urine collection sample. Height, body weight, and percent body fat (seca BIA scale) will be measured. Blood samples will be collected from an antecubital vein with subjects in the seated position by trained phlebotomists. Each blood sample will not exceed 40 ml (2.7 tablespoons). Subjects will also record responses to a 4-week retrospective symptom log. Subjects will be given flavonoid or placebo supplements for the first 4-week period, and ingest the first two supplements in the lab under supervision.

12-WEEK INTERVENTION: Subjects (N=110) will be randomized to the flavonoid supplement or placebo supplement groups for 12 weeks (thus two independent groups run in parallel with 55 subjects). Supplements will be administered in a double-blinded manner, with the code held by Reoxcyn Discoveries Group until the end of the study. The goal is for N=100 subjects to complete all phases of the study. Subjects will ingest two supplement supplements each day of the study, one before breakfast, and the second one before lunch.

Subjects will report to the Human Performance Lab at the 4- and 12-week time points in an overnight-fasted state and repeat all baseline measurements (including the 3-day food record and 24-h urine collection). The 4-week retrospective symptom logs will be filled in at pre-study, 4, 8, and 12 weeks (with the 8-week log administered via email). Subjects will be given an 8-weeks supply of the supplement after completing the 4-week lab session.

SUPPLEMENT INFORMATION:

The flavonoid-rich supplement contains a mixture of flavonoids from green tea and bilberry extracts, and quercetin. The supplement also contains food components that boost flavonoid benefits in the body including fish oil, caffeine, and vitamin C.

The daily dose will be 4 flavonoid tablets (two before breakfast, two before lunch).

Here is a detailed summary of the ingredients of the flavonoid-rich supplement (4 tablets per day):

Supplement Facts Serving size: 4 Tablets Servings per container: 30 Amount per Serving % Daily Value Calories 50 Total Carbohydrate 12 g 4% Sugars 10 g Vitamin C (as Ascorbyl Palmitate) 100 mg 167% Wild Bilberry Fruit Extract (std. min. 25% Total Anthocyanins) 156 mg ** Green Tea Leaf Extract 180 mg ** Quercetin 100 mg ** Natural Caffeine (from Coffea arabica Bean) 100 mg ** NovoOmega® Omega-3 F30 Powder (Std. 30% Omega-3 Fatty Acids (Eicosapentaenoic Acid and Docosahexaenoic Acid)) 200 mg ** * Percent Daily Values are based on a 2,000 calorie diet

** Daily Value not Established Other Ingredients: Sugar, Natural & Artificial Flavor, Dextrose, Cellulose Gum, Sucralose, Bamboo Whole Plant Extract, Guar Gum, Xanthan Gum, Citric Acid, Malic Acid, L-Tartaric Acid Contains Fish.

In general, the flavonoid-rich chewable tablets (4 per day) will provide the equivalent quantity of flavonoids as found in 10 apples, one cup of green tea, and one-fourth cup of bilberries. Consuming 4 tablets per day will add approximately 50% more of the beneficial polyphenols typically consumed by adults.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25 kg/m2 and higher (about 25 pounds or more overweight from recommended levels)
* Generally healthy and without chronic disease including cardiovascular disease (e.g., heart disease, stroke), cancer, type 1 diabetes, rheumatoid arthritis
* Willingness to maintain normal physical activity and diet habits, and make no formal attempts to lose weight during the 12-week study.

Exclusion Criteria:

* Use of Aspirin and non-steroidal anti-inflammatory drugs (NSAIDs) within the past one to two weeks, and plans to use NSAIDs during the 12-week period of the study. Examples include ibuprofen (Advil, Motrin, Nuprin), naproxen (Aleve, Naprosyn), and COX-2 inhibitors (Celebrex).
* Regular use of fish oil supplements, omega 3 supplements, or omega 3-based drugs (Lovaza, etc.) during the past one to two weeks and plans to use these supplements during the study.
* History of allergy or intolerance to green tea, blueberries, fish oil, caffeine, or the flavonoid quercetin.
* Pregnant or breastfeeding
* Currently on a weight reducing plan or using weight-loss medications (e.g., selective serotonin reuptake inhibitors, steroids, Ritalin, appetite suppressors, Xenical, Diethylpropion), and plans to continue during the 12-week period of the study.
* Regular use of large dose nutrient, herbal, and dietary supplements during the past one to two weeks, and plans to use these during the 12-week period of the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Urine phenolics | Change from baseline urine phenolics at 12 weeks
  24-h urine samples collected pre-study and after 12-weeks intervention

SECONDARY OUTCOMES:
Change in global metabolomics | Change from baseline global metabolomics at 12 weeks
  Blood sample analysis for shifts in metabolites pre-study and after 12-weeks intervention
Change in symptoms | Change from baseline symptoms at 4-weeks, 8-weeks, 12-weeks.
  A 4-week retrospective symptom log will be administered pre-study, 4-weeks, 8-weeks, and 12-weeks to document potential adverse gastrointestinal and mental effects.
Change in oxidized LDL | Change from baseline oxidized LDL at 12 weeks
  plasma oxidized LDL
Change in blood diagnostic chemistries | Change from baseline diagnostic chemistries at 12 weeks
  Comprehensive blood diagnostic chemistry panels
Change in CRP | Change from baseline CRP at 12 weeks
  C-reactive protein
Change in IL-6 | Change from baseline IL-6 at 12 weeks
  Plasma IL-6
Change in MCP-1 | Change from baseline MCP-1 at 12 weeks
  Plasma MCP-1
Change in FRAP | Change from baseline FRAP at 12 weeks
  Plasma FRAP

CONTACTS AND LOCATIONS:
Overall Officials: David C Nieman, DrPH, Principal Investigator — Appalachian State Univ
Locations (1):
- Appalachian State University Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through the Human Metabolome Database (HMDB), other public web sites, and publication in the scientific literature.